CLINICAL TRIAL: NCT05809219
Title: The Effect of Different Post-exercise Oral Nutritional Supplement Intake Timing on Sarcopenia Indicators in Hemodialysis Patients
Brief Title: the Effect of Exercise and Oral Supplement Intervention in Sarcopenia Markers in Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Pei-Yu Wu, Project Assistant Professor, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSTC 112-2320-B-039-008
Record Dates: First submitted 2023-03-18; First posted 2023-04-12 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Exercise; Nutritional Status; Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): Participants maintain usual diet and physical activity without any intervention
- 1 hour combined intervention ( Exercise and nutrition) (Experimental): During intervention period, participants have 3 times exercise program per week. Each program is 30 minutes of resistance exercise and aerobic exercise. Participants take oral supplement (103 kcal and 8.4 g of protein) in 1 to 2 hours after exercise program.
  Interventions: Other: 1 hour combined intervention ( Exercise and nutrition)
- 3 hours combined intervention ( Exercise and nutrition) (Experimental): The only one different between "1 hour combined intervention" and this intervention is the time interval between exercise and nutrition. The time interval of "1 hour combined intervention" is 1 to 2 hour, and this intervention is 2.5-4 hours. Other procedure is totally the same.
  Interventions: Other: 3 hours combined intervention ( Exercise and nutrition)
- Nutrition intervention (Experimental): Participants only take oral supplement. The oral supplement is the same as the "1 hour combined intervention" and "3 hours combined intervention".
  Interventions: Dietary Supplement: Nutrition intervention

INTERVENTIONS:
Other: 1 hour combined intervention ( Exercise and nutrition) — Subjects take oral supplement after exercise in the time period between 1-2 hours. They will take oral supplement during hemodialysis treatment.
  Arms: 1 hour combined intervention ( Exercise and nutrition)
Other: 3 hours combined intervention ( Exercise and nutrition) — All procedures between "1 hour combined intervention" and "3 hours combined intervention" are the same. The only one different is the time interval between exercise and nutrition. In this arm, the time interval of exercise and nutrition is 2.5 to 4 hours. When we recruiting subjects, all interventions will be clearly introduced to them, including the same and the different parts among them.
  Arms: 3 hours combined intervention ( Exercise and nutrition)
Dietary Supplement: Nutrition intervention — Subjects only take oral supplement during hemodialysis treatment. The oral supplement is the same as the "1 hour combined intervention" and "3 hours combined intervention".
  Arms: Nutrition intervention

SUMMARY:
Objective: To assess the effect of different post-exercise oral nutritional supplement intake timing on sarcopenia indicators in hemodialysis patients.

Study Design: 24-weeks Randomized Control Trial (RCT), includes 12-wk intervention period and 12-week follow up period.

Setting & Participants: Maintenance hemodialysis patients who were older than 20 years old meet sarcopenia diagnosis criteria.

Intervention: Group A: During intervention period, participants have 3 times exercise program per week. Each program is 30 minutes of resistance exercise and aerobic exercise. Participants take oral supplement in 1 to 2 hours after exercise program. Group B: Participants have the same exercise program and oral supplement as Group A. However, they take oral supplement in 2.5-4 hours after exercise program. Group C: Participants only take oral supplement. Control group: Participants maintain usual diet and physical activity without any intervention.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis treatment longer than 3 months
* Hemodialysis treatment 3 times treatment per weeks
* Kt/V≥1.2 or URR≥65%
* Taking foods by oral
* Meeting the criteria of sarcopenia.

Exclusion Criteria:

* Soy allergy
* Amputation
* Significantly edema
* Receiving palliative care
* Severe angina
* Unstable arrhythmias
* Severe infection
* Heart failure (class 4 of New York Heart Association scale)
* Central venous catheter or femoral arteriovenous fistula
* Pacemaker
* Pregnancy
* Severe paleness
* Severe difficulty breathing
* Chest pain
* Hospitalization 3 months before recruited in this study
* Oral supplement intolerance diagnosed by the doctor or dietitian
* Bone injury/nerve damage/cognition impairment affecting physical activity intervention

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Appendicular skeletal muscle mass | Change from baseline appendicular skeletal muscle mass at 3 months
  The weight of appendicular skeletal muscle mass. This is one of the sarcopenia indicator.
Appendicular skeletal muscle mass | Change from baseline appendicular skeletal muscle mass at 6 months
  The weight of appendicular skeletal muscle mass. This is one of the sarcopenia indicator.
Muscle strength | Change from baseline muscle strength at 3 months
  The measurement of handgrip strength. This is one of the sarcopenia indicator.
Muscle strength | Change from baseline muscle strength at 6 months
  The measurement of handgrip strength. This is one of the sarcopenia indicator.
Physical performance | Change from baseline physical performance at 3 months
  Measuring whether the of 6-meter walk is less than 1.0 m/s or not. This is one of the sarcopenia indicator.
Physical performance | Change from baseline physical performance at 6 months
  Measuring whether the of 6-metre walk is less than 1.0 m/s or not. This is one of the sarcopenia indicator.

CONTACTS AND LOCATIONS:
Overall Officials: PEIYU WU, Principal Investigator — Project Assistant Professor
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
According to the records approved by IRB, the individual participant data of all participants should be protected.